CLINICAL TRIAL: NCT05486351
Title: Keeping Oral o Parental AnticoaguLation in the Acute Phase of Cardioembolic Ischemic
Brief Title: Keeping Oral o Parental AnticoaguLation in the Acute Phase of Cardioembolic Ischemic Stroke
Acronym: KOALA-IS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Hospital Universitario La Paz (Other); Daiichi Sankyo (Industry); Fundación Freno al ICTUS (Unknown)
Responsible Party: Sponsor
Other Study IDs: PI-4056
Record Dates: First submitted 2022-08-02; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Cardioembolic Stroke; Anticoagulant Therapy; Stroke Recurrence; Haemorrhagic Transformation Stroke
MeSH Terms: conditions — Embolic Stroke | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for levels of anticoagulant medications and/or INR testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mantainance of anticoagulation therapy: Patients with acute ischemic stroke of cardioembolic source and previosly anticoagulated in which anticoagulant therapy is mantained
  Interventions: Other: Observation
- Interruption of anticoagulation therapy: Patients with acute ischemic stroke of cardioembolic source and previosly anticoagulated in which anticoagulant therapy is interrupted.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Patients are observed for stroke or systemic embolism and haemorrhagic transformation

SUMMARY:
This is an observational, prospective, multicenter, cohort study in patients with cardioembolic stroke and previous oral or parenteral anticoagulant therapy. Patients in which anticoagulante therapy is mantained will be compared to those in which it is interrupted, in terms of stroke or systemic embolism and haemorrhagic transformation.

DETAILED DESCRIPTION:
Observational, prospective, multicenter, cohort study in patients with recent cardioembolic stroke (<24 hours) and previous oral or parenteral anticoagulant therapy (last dose recieved <24hours) . Patients in which anticoagulante therapy is mantained will be compared to those in which it is interrupted. The decision to mantain or interrumpt the anticoagulant therapy is made by the treating physician as hospital protocol. Stroke recurrence, haemorrhagic transformation at 90 days are evalauted and also complication during the hospitalization and functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke of less than 24 hours since beginning of symptoms or last seen normal
* Mayor cardioembolic source (atrial fibrilation or flutter, mechanical heart valve prosthesis, recient miocardic infarction, rheumatic mitral valve stenosis, dilated cardiomyopathy, atrial myxoma, left ventricular focal akynesia.
* Previous treatment with oral anticoagulants (vitamin K antagonists or direct oral anticoagulants), having received the last dose within the previous 24 hours. Treatment with intravenous or subcutaneos heparin is also valid.
* Age >18 years-old
* Signed informed consent (by patient or representative)

Exclusion Criteria:

* History of Intracraneal or extracraneal haemorrhage that contraindicates anticoagulant therapy
* Patients treated with intravenous thrombolysis as a reperfusion therapy
* Intracraneal haemorrhage on initial CT scan
* Health status with a short survival prevision
* Patients in which a neurosurgery intervention could be indicated
* Child-bearing woman or in breast-feeding period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke, with a major cardioembolic source and previosly treated with oral or parental anticoagulants.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Ischemic stroke recurrence | 90 days
  recurrence of ischemic stroke noticied by changes in neurologic status and supported by neuroimaging
Symptomatic haemorrhagic transformation | 90 days
  Symptomatic haemorrhagic transformation defined by the SITS criteria and supported by neuroimaging

SECONDARY OUTCOMES:
Early ischemic stroke recurrence | Day 1 or day 7
  Recurrence of ischemic stroke at days 1 or day 7
Early symptomatic haemorrhagic transformation | Day 1 or day 7
  Symptomatic transformation ocurring on day 1 or day 7
Early radiologic haemorrhagic transformation | Day 1 or day 7
  Parenchymal haematoma (type PH1 or PH2) on control neuroimaging performed at 24h (if mechanical thromectomy performed) and at day 7
Systemic embolism | Day 1, day 7 or day 90
  Clinical, radiologic or analytic findings that suggest an ischemic event (myocardic, renal, splenic, bowl or limb infarctions
Major extracraneal haemorrhagic complication | Day 1, day 7 or day 90
  intraocular, intraspinal, pericardic, intra-articular, intra-muscular with compartimental syndrome, retro-peritoneal bleeding that requires surgery or that causes death. Definition according to ISTH criteria
Mortality | Day 7
  Death
Neurologic status | Day 90
  NIHSS scale
Functional status | Day 90
  modified Rankin scale

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Rigual Bobillo, MD, Principal Investigator — Hospital Universitario La Paz
Locations (3):
- Bichat Claude Bernard Hospital, Paris, France
- Spain (2):
  - Jimenez Diaz Fundation University Hospital, Madrid
  - La Paz University Hospital, Madrid

IPD SHARING:
Plan to Share IPD: Undecided